CLINICAL TRIAL: NCT04063644
Title: Effect of Visglyc on the Quality of Life of Patients With Dry Eye Symptomatology and Age-related Loss of Visual Acuity
Brief Title: Quality of Life and Visual Acuity of Visglyc Eye Drops on Dry Eye Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: OPKO Health, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: OPK-GLY-2018-01
Record Dates: First submitted 2019-08-13; First posted 2019-08-21 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Dry Eye Syndromes; Cataract
Keywords: Dry eye; Cataract; Visual acuity; Quality of life; Eye drops; Dry eye symptomatology; N-acetylcarnosine; Vaccinium myrtillus; Chondroitin sulfate; Chondroitin sulphate; N-Acetylcharnosine
MeSH Terms: conditions — Dry Eye Syndromes; Cataract

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single-blinded: The physician performing the recruiting will be different and cannot be related to the investigator evaluating the follow-up.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vis Glyc Neo (Experimental): Vis glyc eye drops is administered.
  Eye drops based on N-Acetylcoarnosine, Vaccinium myrtillus and Chondroitin sulfate
  Interventions: Device: Vis Glyc Neo
- physiological saline solution (Active Comparator): Physiological saline solution ALVITA is administered.
  Interventions: Device: Physiological saline solution

INTERVENTIONS:
Device: Vis Glyc Neo — 1 drop in each eye, three times a day.
  Arms: Vis Glyc Neo
Device: Physiological saline solution — 1 drop in each eye, three times a day.
  Arms: physiological saline solution

SUMMARY:
Clinical trial with medical devices, post-authorization, parallel, single-blind, randomized, comparative, prospective to study how afects the quality of life the use of ocular eye drops on patients with dry eye symptomatology and age-related loss of visual acuity.

Secondary purposes: efects on the dry eye symptomatology, efect on visual acuity and treatment adherence.

ELIGIBILITY:
Inclusion Criteria:

* Subjects between the ages of 50 and 70.
* Subjects with initial or slight changes characteristic of cataracts (grade 1-3 according to LOCS III classification).
* Subjects with dry eye symptoms.
* Confirmation of senile cataract diagnosis according to medical history and clinical observations, bilateral.
* Visual acuity equal to or greater than (0.6) in both eyes (with the best correction).
* Cataracts without the need for surgical intervention in the near future (1 year) based on the visual needs of the patient and ocular symptomatology.
* Subjects that have not undergone cataract surgery.
* Cases that do not accept surgery (weak corneas, high degree of myopia, sensitivity to light, severe dryness of the eyes or by their own decision).
* Subjects who agree to sign the IC (Informed Consent).

Exclusion Criteria:

* Subjects with eye diseases such as glaucoma or diabetic retinopathy.
* Previous laser photocoagulation of the retina.
* Previous corneal or anterior segment surgery or previous corneal scars that may interfere with visualization or photographs.
* Presence of mature cataracts (grade 4-5/6 according to LOCS III classification) in both eyes.
* Candidates for surgery in the following year.
* Subjects with monocular aphakia (absence of crystalline lens) or secondary cataracts (associated with steroid use, local or total irradiation, local inflammation or degenerative processes, ocular trauma).
* Subjects with known hypersensitivity to any component of ophthalmic treatment.
* Subjects treated with drugs that may interfere with the evolution of the disease under study.
* Subjects who wear contact lenses.
* Pregnant women.
* Breastfeeding women.
* Subjects who have participated in another clinical trial within the last 30 days.
* Subjects with linguistic or psychological incapacity to understand and sign the CI.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2019-05-30 (Actual); Primary Completion 2020-12-22 (Actual); Study Completion 2020-12-22 (Actual)

PRIMARY OUTCOMES:
Change in quality of visual life: NEI VFQ-25 questionnaire | Change from baseline quality of life at 6 months
  In patients with dry eye symptomatology and age-related loss of visual acuity. Assessed using NEI VFQ-25 questionnaire. It is a questionnaire with 25 questions.
  Its format is divided into 4 subscales: visual function, difficulty with activities, driving a car and responding to vision problems. It consists of a base of 25 questions (each with five or six levels of response and scoring ranges) addressed to vision, representing 11 domains, elements or items related to health; 1) general vision, 2) eye pain, 3) near activities, 4) distance activities, 5) social functioning, 6) mental health, 7) role difficulties or limitations, 8) dependence, 9) driving, 10) color vision and 11) peripheral vision.
  Each domain receives an evaluation from 0 to 100; the high evaluation represents changes in visual functioning, where 0 is the lowest and 100 is the best possible.

SECONDARY OUTCOMES:
Change in quality of visual life: NEI VFQ-25 questionnaire | 0, 30, 90, 180 days
  In patients with dry eye symptomatology and age-related loss of visual acuity. Assessed using NEI VFQ-25 questionnaire. It is a questionnaire with 25 questions.
  Its format is divided into 4 subscales: visual function, difficulty with activities, driving a car and responding to vision problems. It consists of a base of 25 questions (each with five or six levels of response and scoring ranges) addressed to vision, representing 11 domains, elements or items related to health; 1) general vision, 2) eye pain, 3) near activities, 4) distance activities, 5) social functioning, 6) mental health, 7) role difficulties or limitations, 8) dependence, 9) driving, 10) color vision and 11) peripheral vision.
  Each domain receives an evaluation from 0 to 100; the high evaluation represents changes in visual functioning, where 0 is the lowest and 100 is the best possible.
Visual Acuity Evaluation I | 0, 90, 180 days
  To assess the age-related visual acuity in patients.
  - The CSV-1000E contrast sensitivity test. This test provides for four (4) rows of sine-wave gratings. These gratings test the spatial frequencies of 3, 6, 12 and 18 cycles/degree (CPD). The levels of contrast are 1 to 8. The higher the contrast or modulation, the greater the difference in luminance and the better the object will be distinguished from the background.
Visual Acuity Evaluation II | 0, 90, 180 days
  To assess the age-related visual acuity in patients.
  - LOCS III classification of cataract grade using images obtained by ophthalmoscopy with slit lamp, which allows the study of the anterior segment of the patient's eye. It consists of six slit lamp images to evaluate core color (NC) and opalescence (NO); five backlit images to evaluate cortical cataract (C); and five backlit images to evaluate posterior subcapsular cataract (P). The severity of the cataract is classified on a decimal scale, and the patterns have regularly separated intervals on a decimal scale.
Visual Acuity Evaluation III | 0, 90, 180 days
  To assess the age-related visual acuity in patients.
  - Visual acuity test with the best correction in each eye using Snellen E-screens, measured in decimal system and MAR logarithm. Level of vision with respect to the row in Snellen's graph, which the rows consist of 1 to 11. The lower the row (greater numbers) the patient can distinguish, the greater the visual acuity he will have.
Dry eye symptomatology Evaluation I | 0, 90, 180 days
  Schirmer I test (without anesthesia): to determine the dryness of the eye. It consists of placing a thin strip of paper at the bottom of the conjunctival sac and before this foreign body see the patient's tear production capacity (measuring the wet area in mm). The less mm the less tear production capacity.
Dry eye symptomatology Evaluation II | 0, 90, 180 days
  - Fluorescein staining test: to assess dryness of the eye. Fluorescein is instilled in both conjunctival sacs. Absence of staining indicates integrity of the corneal epithelium. There are degrees of fluorescein staining from 0 to 5. The highest the worst results.
Dry eye symptomatology Evaluation III | 0 and 180 days
  The OSDI Test (ocular surface disease index) is a simple test created to establish the severity and classification of dry eye according to its symptoms. It is based on 12 different questions about situations related to patient symptomatology.
  A score of 100 corresponds to a total disability (answer "At all times" to all questions answered), while a score of 0 corresponds to no disability.
Treatment adherence | 30, 90 and 180 days
  Ask patients about the daily administration of the treatment according to the protocol.
Adverse events | 30, 90 and 180 days
  Number of participants with Adverse events and types of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Beatriz Sarmiento Torres, MD, MSc, Principal Investigator — Hospital Universitario 12 Octubre
Locations (1):
- Hospital Universitario 12 de Octubre, Madrid, Spain

IPD SHARING:
Plan to Share IPD: No